CLINICAL TRIAL: NCT02999854
Title: A Phase III, Multicenter, Randomized Controlled Study to Compare Safety and Efficacy of a Haploidentical HSCT and Adjunctive Treatment With ATIR101, a T-lymphocyte Enriched Leukocyte Preparation Depleted ex Vivo of Host Alloreactive T-cells, Versus a Haploidentical HSCT With Post-transplant Cyclophosphamide in Patients With a Hematologic Malignancy
Brief Title: Safety and Efficacy of ATIR101 as Adjunctive Treatment to Blood Stem Cell Transplantation From a Haploidentical Family Donor Compared to Post-transplant Cyclophosphamide in Patients With Blood Cancer
Acronym: HATCY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient efficacy, terminated by Sponsor
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR-AIR-009; 2016-004672-21 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: Haploidentical stem cell transplantation; Graft-versus-host disease; Immune reconstitution; Alloreactive T-cells; Photodynamic treatment; Hematologic malignancy; Transplant-related mortality; Overall survival; GRFS; GVHD
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Graft vs Host Disease; Hematologic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATIR101 (Experimental): T-cell depleted HSCT from a related, haploidentical donor, followed by IV infusion with ATIR101 at a single dose of 2×10E6 viable T-cells/kg body weight between 28 and 32 days after the HSCT
  Interventions: Biological: ATIR101; Procedure: T-cell depleted HSCT from a related, haploidentical donor
- PTCy (Active Comparator): T-cell replete HSCT from a related, haploidentical donor, followed by IV infusion of post-transplant cyclophosphamide (PTCy) 50 mg/kg/day at 3 and 4/5 days after the HSCT
  Interventions: Drug: Cyclophosphamide; Procedure: T-cell replete HSCT from a related, haploidentical donor

INTERVENTIONS:
Biological: ATIR101 — ATIR101 is a T-lymphocyte enriched leukocyte preparation depleted ex vivo of host alloreactive T-cells using photodynamic treatment; single dose of 2×10E6 viable T-cells/kg body weight between 28 and 32 days after the HSCT (intravenous infusion)
  Arms: ATIR101
Drug: Cyclophosphamide — High dose post-transplant cyclophosphamide 50 mg/kg/day at 3 and 4/5 days after the HSCT (powder for intravenous infusion)
  Arms: PTCy
Procedure: T-cell depleted HSCT from a related, haploidentical donor — T-cell depleted graft prepared from peripheral blood stem cells using the CD34+ cell selection method; infused after a total body irradiation (TBI) or non-TBI conditioning regimen
  Arms: ATIR101
Procedure: T-cell replete HSCT from a related, haploidentical donor — T-cell replete (full, non-manipulated) graft prepared from either bone marrow or peripheral blood stem cells; infused after a total body irradiation (TBI) or non-TBI conditioning regimen
  Arms: PTCy

SUMMARY:
The primary objective of this study is to compare safety and efficacy of a haploidentical T-cell depleted HSCT and adjunctive treatment with ATIR101 versus a haploidentical T cell replete HSCT with post-transplant administration of high dose cyclophosphamide (PTCy) in patients with a hematologic malignancy. An additional objective of the study is to compare the effect of the two treatments on quality of life.

DETAILED DESCRIPTION:
Study CR-AIR-009 is a Phase III randomized controlled multicenter open-label study comparing two parallel groups. After signing informed consent, a total of 250 patients will be randomized in a 1:1 fashion to receive either a T-cell depleted hematopoietic stem cell transplantation (HSCT; CD34 selection) from a related, haploidentical donor, followed by ATIR101 infusion, or a T-cell replete HSCT, followed by a high dose of post-transplant cyclophosphamide (PTCy).

Randomization will use minimization to balance treatment groups with respect to underlying disease (AML, ALL, or MDS), Disease Risk Index (DRI; intermediate risk, high risk, or very high risk) and center. A stochastic treatment allocation procedure will be used so that the treatment assignment is random for all patients entered in the study.

Patients randomized in the ATIR101 group will receive a single ATIR101 dose of 2×10E6 viable T-cells/kg between 28 and 32 days after the HSCT. Patients randomized in the PTCy group will receive cyclophosphamide 50 mg/kg/day at 3 and 4/5 days after the HSCT. All patients will be followed up for at least 24 months post HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following hematologic malignancies:

  * Acute myeloid leukemia (AML) in first cytomorphological remission (with < 5% blasts in the bone marrow) with Disease Risk Index (DRI) intermediate or above, or in second or higher cytomorphological remission (with < 5% blasts in the bone marrow)
  * Acute lymphoblastic leukemia (ALL) in first or higher remission (with < 5% blasts in the bone marrow)
  * Myelodysplastic syndrome (MDS): transfusion-dependent (requiring at least one transfusion per month), or intermediate or higher Revised International Prognostic Scoring System (IPSS-R) risk group
* Clinical justification of allogeneic stem cell transplantation where a suitable HLA matched sibling or unrelated donor is unavailable in a timely manner
* Availability of a related haploidentical donor with one fully shared haplotype and 2 to 4 mismatches at the HLA-A, -B, -C, and -DRB1 loci of the unshared haplotype, as determined by high resolution human leukocyte antigen (HLA)-typing
* Karnofsky Performance Status (KPS) ≥ 70%
* Male or female, age ≥ 18 years and ≤ 70 years. Patients aged ≥ 65 years must have a Sorror score ≤ 3
* Patient weight ≥ 25 kg and ≤ 130 kg
* Availability of a donor aged ≥ 16 years and ≤ 75 years who is eligible according to local requirements and regulations. Donors aged < 16 years are allowed if they are the only option for an HSCT, if they are permitted by local regulations, and if the IRB/IEC approves participation in the study.
* For females of childbearing potential who are sexually active and males who have sexual contact with a female of childbearing potential: willingness to use of reliable methods of contraception (oral contraceptives, intrauterine device, hormone implants, contraceptive injection or abstinence) during study participation
* Given written informed consent (patient and donor)

Exclusion Criteria:

* Diagnosis of chronic myelomonocytic leukemia (CMML)
* Availability of a suitable HLA-matched sibling or unrelated donor in a donor search
* Prior allogeneic hematopoietic stem cell transplantation
* Diffusing capacity for carbon monoxide (hemoglobin corrected DLCO) < 50% predicted
* Left ventricular ejection fraction < 45% (evaluated by echocardiogram or MUGA scan)
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (CTCAE grade 2)
* Creatinine clearance < 50 ml/min (calculated or measured)
* Positive pregnancy test or breastfeeding of patient or donor (women of childbearing age only)
* Estimated probability of surviving less than 3 months
* Known allergy to any of the components of ATIR101 (e.g., dimethyl sulfoxide)
* Known hypersensitivity to cyclophosphamide or any of its metabolites
* Any contraindication for GVHD prophylaxis with mycophenolate mofetil, cyclosporine A, or tacrolimus
* Known presence of HLA antibodies against the non-shared donor haplotype
* Positive viral test of the patient or donor for human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B virus (HBV), hepatitis C virus (HCV), Treponema pallidum, human T-lymphotropic virus (HTLV)-1 (if tested), HTLV-2 (if tested), West Nile virus (WNV; if tested), or Zika virus (if tested)
* Any other condition that, in the opinion of the investigator, makes the patient or donor ineligible for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Claude Roy, Prof MD, Principal Investigator — Research Center and Cellular Therapy Laboratory, Maisonneuve-Rosemont Hospital (Montreal, Canada); Stephan Mielke, Prof MD, Principal Investigator — Centre for Allogeneic Stem Cell Transplantation, Karolinska University Hospital (Stockholm, Sweden)
Locations (42):
- United States (12):
  - City of Hope National Medical Center, Duarte, California
  - Moores UC San Diego Cancer Center, La Jolla, California
  - UCLA Center for Health Sciences, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Emory University, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Oregon Health & Science University, Portland, Oregon
- Belgium (5):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada
- University Hospital Centre Zagreb, Zagreb, Croatia
- APHP Hospital Saint Louis, Paris, France
- Germany (4):
  - University Hospital Frankfurt, Goethe University, Frankfurt
  - University Medical Center Mainz, Mainz
  - Ludwig-Maximilians-University Hospital of Munich-Grosshadern, Munich
  - Universitätsklinikum Würzburg, Würzburg
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center & Hadassah Hospital Ein Karem, Jerusalem
  - Sourasky Medical Center & Tel Aviv University, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (2):
  - Milano Hospital, Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Faculdade de Medicina da Universidade de Lisboa, Lisbon, Portugal
- Spain (4):
  - University Hospital Barcelona Vall d' Hebron, Barcelona
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - UGC Hematología y Hemoterapia, Seville
  - Servicio de Hematología Hospital, Universitari I politècnic La Fe, Valencia
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (5):
  - Heartlands Hospital, Birmingham
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Hammersmith Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Active Study Phase (up to 18 Months)
Arm/Group | ATIR101 | PTCy
Started | 32 | 31
Completed | 8 | 22
Not Completed | 24 | 9
Not completed — Screen failures | 7 | 2
Not completed — Discontinued before HSCT | 8 | 2
Not completed — Death | 7 | 5
Not completed — Completed 2 year follow-up | 1 | 0
Not completed — End of study after HSCT but before treatment | 1 | 0
Period: Long Term Safety FU (up to 24 Months)
Arm/Group | ATIR101 | PTCy
Started | 8 | 22
Completed | 5 | 19
Not Completed | 3 | 3
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATIR101 | PTCy | Total
Number analyzed (Participants) | 16 | 27 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.63) | 32.8 (13.20) | 34.5 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 12 | 22 | 34
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 23 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Hematologic malignancy [Count of Participants; unit: Participants]
  Acute lymphatic leukemia (ALL) | 4 | 2 | 6
  Acute myeloid leukemia (AML) | 9 | 18 | 27
  Myelodysplastic syndrome (MDS) | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Graft-versus-host Disease-free, Relapse-free Survival (GRFS)
Description: Defined as the time until acute GVHD grade III/IV, chronic GVHD requiring systemic treatment, relapse, or death, whichever occurs first. Kaplan-Meier estimates (percentage of participants) of GRFS were calculated at 24 months post HSCT.
Time Frame: 24 months post-HSCT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 16 | 27
Percentage of participants | 25 [8 to 47] | 62 [41 to 78]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from HSCT until death from any cause. Kaplan-Meier estimates (percentage of participants) of OS were calculated at 24 months post HSCT.
Time Frame: 24 months post-HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 16 | 27
percentage of participants | 49 [24 to 71] | 77 [55 to 89]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from HSCT until relapse, disease progression, or death, whichever occurs first. Kaplan-Meier estimates (percentage of participants) of PFS were calculated at 24 months post HSCT.
Time Frame: 24 months post-HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 16 | 27
percentage of participants | 44 [20 to 66] | 73 [52 to 86]

4. Secondary Outcome: Relapse-related Mortality (RRM)
Description: Time from randomization to death due to disease relapse or disease progression
Time Frame: Through study completion, at least two years post HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Transplant-related Mortality (TRM)
Description: Defined as death due to causes other than disease relapse or progression, or other causes which are unrelated to the transplantation procedure (e.g. accident, suicide). Kaplan-Meier estimates (percentage of participants) of PFS were calculated at 24 months post HSCT.
Time Frame: 24 months post-HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 16 | 27
percentage of participants | 44 [19 to 66] | 15 [5 to 31]

6. Other Pre Specified Outcome: Immune Reconstitution
Description: Time to CD3+ > 0.2×10E9/l in peripheral blood (at two consecutive measurements; time to first measurement)
Time Frame: Through study completion, at least two years post HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Cumulative Incidence of Grade II-IV and Grade III-IV Acute Graft-versus-host-disease (GVHD)
Time Frame: Through study completion, at least two years post HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Cumulative Incidence of Moderate/Severe Chronic GVHD
Time Frame: Through study completion, at least two years post HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Cumulative Incidence of Chronic GVHD Requiring Systemic Immunosuppressive Treatment
Time Frame: Through study completion, at least two years post HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Duration of GVHD Episodes
Time Frame: Through study completion, at least two years post HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Cumulative Incidence of NCI CTCAE Grade 2-5 and Grade 3-5 Infections
Description: Viral, fungal, and bacterial infections
Time Frame: Until 2 years after the HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Cumulative Incidence of NCI CTCAE Grade 3-5 Adverse Events
Description: Viral, fungal, and bacterial infections
Time Frame: Until 2 years after the HSCT
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: FACT-BMT Total Score (Change From Screening)
Description: Quality of life: Foundation for the Accreditation of Cellular Therapy - Bone Marrow Transplantation questionnaire (FACT-BMT)
Time Frame: Through study completion (Month 3, 6, 12, 24, 36, 48 post HSCT)
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: SF-36 Total Score (Change From Screening)
Description: Quality of life: Short Form 36-item health survey (SF-36)
Time Frame: Through study completion (Month 3, 6, 12, 24, 36, 48 post HSCT)
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: MDASI Total Score (Change From Screening)
Description: Quality of life: MD Anderson Symptom Inventory (MDASI)
Time Frame: Through study completion (Month 3, 6, 12, 24, 36, 48 post HSCT)
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: EQ-5D-5L (Change From Screening)
Description: Quality of life: EQ-5D-5L
Time Frame: Through study completion (Month 3, 6, 12, 24, 36, 48 post HSCT)
Population: Study was pre-maturely terminated. Data not collected.
Arm/Group | ATIR101 | PTCy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Long term safety follow-up, 24 months.
Description: Study was pre-maturely terminated. For the long term safety follow-up (LTFU), up to 24 months post-HSCT, only cumulative SAEs were recorded.
  (63 patients had been enrolled (randomized); 32 to ATIR101 group and 31 to PTCy group (intention-to-treat [ITT] population). Only patients who received an HSCT and ATIR101 (n=16) or at least one dose of PTCy (n=27) were included in the modified ITT population (MITT). Eight ATIR101, and 22 PTCy treated patients entered 2 year LTFU).
Arm/Group | ATIR101 | PTCy
All-Cause Mortality (participants affected / at risk) | 8/16 | 6/27
Serious Adverse Events (participants affected / at risk) | 13/16 | 19/27
Other Adverse Events (participants affected / at risk) | 0/16 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATIR101 (N=16) | PTCy (N=27)
Infections and infestations (Infections and infestations) | 10 | 12
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 | 5
General disorders and administration site conditions (General disorders) | 4 | 6
Cardiac disorders (Cardiac disorders) | 2 | 5
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 3
Nervous system disorders (Nervous system disorders) | 3 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 | 0
Investigations (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT02999854/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT02999854/SAP_001.pdf